CLINICAL TRIAL: NCT07285330
Title: NUTRI-DIAB: Impact of the Dietitian-Nutritionist Model vs. Day Hospital on the Metabolic Control of Patients With Type 2 Diabetes
Brief Title: Dietitian-Nutritionist vs. Day Hospital in the Metabolic Control of Patients With Type 2 Diabetes
Acronym: NUTRI-DIAB
Status: Recruiting | Type: Observational
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Other Study IDs: CSAPG-76
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Diabetes (DM)
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Nutritionists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Day Care Hospital: These patients received joint care from a nurse and an endocrinologist in the day hospital before 2024.
  Interventions: Other: Day Care Hospital
- Nutritionist: These patients received joint care from a nutriotinist and finally an endocrinologist in ambulatory care unit after 2024.
  Interventions: Other: Nutritionist

INTERVENTIONS:
Other: Day Care Hospital — Clinical follow-up under the joint care of a nurse and an endocrinologist at Day Care Hospital
  Groups: Day Care Hospital
Other: Nutritionist — Clinical follow-up with a dietitian-nutritionist and an endocrinologist at ambulatory care unit
  Groups: Nutritionist

SUMMARY:
The present study aims to compare the effects on glycated hemoglobin (HbA1c) at 3 months of two care models in patients with type 2 diabetes referred due to poor glycemic control: a day hospital endocrinology care model versus a care model centered on follow-up by a dietitian-nutritionist.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of type 2 diabetes (T2DM) referred to endocrinology due to poor metabolic control.
* Patients on insulin therapy

Exclusion Criteria:

* Referred from primary care for other reasons such as hypoglycemia.
* Patients with other types of diabetes mellitus or with uncertainty in diagnostic classification.
* Patients on rapid-acting insulin bolus therapy.
* Patients with acute decompensation of diabetes.
* Patients receiving corticosteroid treatment.
* Dependent individuals for activities of daily living (ADL) with a Barthel index score below 60 or with cognitive impairment.
* Language barrier.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by diabetes mellitus type 2
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Glycate hemoglobin | three months after completion of the intervention
  Glycated hemoglobin (HbA1c) levels three months after completion of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Vilafranca, Vilafranca del Penedès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.